CLINICAL TRIAL: NCT03917810
Title: Acute Responses to Manipulating Dietary Carbohydrate Content on Free-living Physical Activity Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Senior Lecturer, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP 17/18 219
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Physical Activity
Keywords: Nutrition; Carbohydrates; Ketogenic; Metabolism
MeSH Terms: conditions — Motor Activity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomised crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MODSUG (Active Comparator): Diet consisting of 50% carbohydrate (20% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOWSUG (Experimental): Diet consisting of 50% carbohydrate (<5% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOWCHO (Experimental): Diet consisting of <8% carbohydrate (<5% sugar), 15% protein, >77% fat
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Macronutrient composition (specifically type and/or amount of carbohydrate) is manipulated

SUMMARY:
Dietary sugar and carbohydrate intakes will be manipulated for 3 days in a randomised crossover design. All food will be provided. Free-living physical activity energy expenditure will be measured using combined heart rate and accelerometry. Metabolic and appetite/mood responses to 3 days on each diet will be measured.

Each participant will undergo 3 days of each diet:

1. Moderate sugar - reflecting the composition of a typical European diet
2. Low sugar - similar macronutrient composition of a typical European diet but with <5% energy intake from free sugars (as per government guidelines)
3. Low carbohydrate - low carbohydrate diet with <5% energy intake from sugar and <8% energy intake from carbohydrate, replacing carbohydrate energy with fat

DETAILED DESCRIPTION:
Guidelines calling for dietary free sugars to be reduced have been formulated from evidence that diets high in sugar are associated with high energy intake. In theory, by reducing the intake of sugars, calorie surplus will be reduced and energy balance will be maintained. However, when referring to interventions/behaviours that influence energy balance, both sides of the energy balance equation need to be considered. Alterations in nutrients may influence aspects of energy expenditure, not solely energy intake, and this may have implications for the efficacy of guidelines seeking to influence energy intake.

It is important to consider energy expenditure in the context of health. The most variable component of energy expenditure between individuals is physical activity energy expenditure (PAEE), which varies from ~600-2100 kcal per day in men of a similar demographic. Current guidelines do not regard the effect that changing dietary sugar might have on PAEE and therefore total energy expenditure.

Furthermore, there is increasing interest in restricting overall carbohydrate intake to treat metabolic disease or achieve ketogenesis. Very little is known about nutrition-physical activity interactions with this type of intervention.

This study will prescribe 3 diets to healthy males for 3 days in a randomised crossover design, where each participant will consume each of the diets. All food will be prepared and provided by the study team. The diets are as follows:

1. Moderate sugar - reflecting the composition of a typical European diet
2. Low sugar - similar macronutrient composition of a typical European diet but with <5% energy intake from free sugars (as per government guidelines)
3. Low carbohydrate - low carbohydrate diet with <5% energy intake from sugar and <8% energy intake from carbohydrate, replacing carbohydrate energy with fat

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-29.9 kg∙m-2
* Age 18-65 years
* Male
* Able and willing to provide informed consent and safely comply with study procedures
* No anticipated changes in physical activity during the study (e.g. holidays)

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)•Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (±3%)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Physical activity energy expenditure (kj/day or kcal/day) | 3 days
  Physical activity energy expenditure measured using individually-calibrated combined heart rate and accelerometry (kj/day or kcal/day)

SECONDARY OUTCOMES:
Time spent in different physical activity intensities (MET categories) (minutes) | 3 days
  Time spent in different physical activity intensities (MET categories) (minutes) using individually-calibrated combined heart rate and accelerometry
Energy expended in different physical activity intensities (MET categories) (kJ/day or kcal/day) | 3 days
  Energy expended in different physical activity intensities (MET categories) (kJ/day or kcal/day) using individually-calibrated combined heart rate and accelerometry
Energy expended in the postprandial period (kJ or kcal) | 3 days
  Energy expended in the postprandial period (kJ or kcal) measured using individually-calibrated combined heart rate and accelerometry
Fasting blood glucose concentrations | 3 days
  Measures of blood glucose concentrations pre- and post-intervention.
Fasting blood insulin concentrations | 3 days
  Measures of blood insulin concentrations pre- and post-intervention.
Fasting blood triglyceride concentrations | 3 days
  Measures of blood triglyceride concentrations pre- and post-intervention.
Fasting blood non-esterified fatty acid concentrations | 3 days
  Measures of blood non-esterified fatty acid concentrations pre- and post-intervention.
Fasting blood lactate concentrations | 3 days
  Measures of blood lactate concentrations pre- and post-intervention.
Fasting blood beta-hydroxybutyrate concentrations | 3 days
  Measures of blood beta-hydroxybutyrate concentrations pre- and post-intervention.
Fasting blood leptin concentrations | 3 days
  Measures of blood leptin concentrations pre- and post-intervention.
Fasting blood fibroblast growth factor-21 concentrations | 3 days
  Measures of blood fibroblast growth factor-21 concentrations pre- and post-intervention.
Fasting blood total cholesterol concentrations | 3 days
  Measures of blood total cholesterol concentrations pre- and post-intervention.
Fasting blood high density lipoprotein concentrations | 3 days
  Measures of blood high density lipoprotein concentrations pre- and post-intervention.
Fasting blood low density lipoprotein concentrations | 3 days
  Measures of blood low density lipoprotein concentrations pre- and post-intervention.
Food preference ratings | 3 days
  Food preference ratings determined by computer task measured pre- and post-intervention
Subjective appetite and mood ratings | 3 days
  Measured by 0-100 mm visual analogue scales measured pre- and post-intervention
Blood pressure | 3 days
  Blood pressure using an automated sphygmomanometer pre- and post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

REFERENCES:
- [Background] Smith HA, Gonzalez JT, Thompson D, Betts JA. Dietary carbohydrates, components of energy balance, and associated health outcomes. Nutr Rev. 2017 Oct 1;75(10):783-797. doi: 10.1093/nutrit/nux045. PMID 29028272
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233